CLINICAL TRIAL: NCT04275791
Title: Assessment of the Benefit of an Inclusive Health Organization on the Prognosis of Severe Trauma Patients
Acronym: TRAUMINXCLUSIF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: APHP180625
Record Dates: First submitted 2020-01-31; First posted 2020-02-19 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Wounds and Injuries
Keywords: Advanced Trauma Life Support Care; Trauma Severity Indices; Trauma Centers; Triage
MeSH Terms: conditions — Wounds and Injuries | interventions — Triage

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hierarchized (Experimental): Structured regional health organization, composed of trauma centers hierarchized in several levels according to their capacity to receive severe traumatized persons.
  Interventions: Other: Triage
- all-or-nothing (No Intervention): Structured regional health organization, composed of non-hierarchical trauma centers at different levels according to their capacity to receive severe trauma victims (all-or-nothing type).

INTERVENTIONS:
Other: Triage — Experimental : Trauma patient orientation in a structured regional health organization, composed of trauma centers hierarchized in several levels according to their capacity to receive severe traumatized persons.
  Arms: hierarchized

SUMMARY:
Appropriate management reduces the mortality of severe trauma victims. This is based on a pre-hospital medical assessment of severity, the initiation of life-saving treatments at the pre-hospital level, and referral to a hospital with human and material resources adapted to the patient's severity. The objective of this research project is to show that the 28-day mortality after severe trauma is lower in a structured health system, compared to a non-structured system.

DETAILED DESCRIPTION:
Appropriate management reduces the mortality of severe trauma victims defined by an Injury Severity Score (ISS) greater than 15 or the need for specialized and/or urgent treatment. This is based on a pre-hospital medical assessment of severity, the initiation of life-saving treatments at the pre-hospital level, and referral to a hospital with human and material resources adapted to the patient's severity.

The trauma hospital organisation in France is of the "exclusive" type. It contrasts trauma centres with other hospitals, only providing care for severe trauma victims in the former, which are most often confused with university hospitals. The choice of referral to this type of centre is made using a triage algorithm known as "de Vittel". In addition to an insufficient network within a region leading to longer hospital access time, this organisation leads to saturation of the referral centres by patients with few lesions. For this reason, this organisation has been rethought in an innovative way within the Auvergne-Rhône-Alpes region, in favour of an "inclusive" system that takes the form of a network of hospitals with capacities to receive severely traumatised patients that vary according to their equipment and personnel. Patients are referred within this network according to their severity category (unstable, stabilized or stable).

The main objective is to show that the 28-day mortality of severely traumatized persons oriented according to their severity in an inclusive system is lower, at identical severity, than in a conventional exclusive system in which the orientation is guided by the Vittel algorithm.

Secondary objectives are to show that the management of severe traumatized persons oriented according to their severity in an inclusive system, compared to the management in an exclusive conventional system in which the orientation is guided by the Vittel/ASCOTT algorithm, is associated, at identical severity, with :

* Less under-triage;
* Less over-triage;
* A lower incidence of secondary transfers to a trauma center;
* A greater number of days living without mechanical ventilation (during the first 28 days);
* More days living without resuscitation (within the first 28 days);
* More frequent and rapid use of whole-body CT scans with contrast injection;
* More frequent and rapid use of specialized emergency therapies (laparotomy or hemostasis thoracotomy, embolization, craniectomy, intracranial pressure measurement, chest drainage).

ELIGIBILITY:
Inclusion Criteria:

- Patients cared for in the aftermath of a severe trauma, by a pre-hospital medical team regulated by the territorially competent SAMU, who arrived at the hospital alive.

Exclusion Criteria:

* Age < 18 years
* Patients with no signs of life on hospital arrival and reported deceased within 30 minutes of admission
* Patients with severe burns (>10% skin area burned)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
28-day mortality | 28th day
  The primary endpoint will be 28-day mortality, defined as the occurrence of death from any cause within the first 28 days following trauma.

SECONDARY OUTCOMES:
Undertriage | 28th day
  Undertriage, defined as the management outside the trauma care system adapted to their condition of patients whose ISS is strictly greater than 15, or presenting at least one of the following criteria:
  * the need for transfusion of more than 4 red blood cell concentrates during the first 6 hours of management;
  * the presence of severe head trauma with CT scan lesions;
  * the presence of a spinal cord injury;
  * the need for specialized emergency surgery (laparotomy or hemostasis thoracotomy, embolization, craniectomy, intracranial pressure measurement, chest drainage) within the first 24 hours;
  * the need for a secondary inter-hospital transfer to a trauma center. This variable will be assessed at the end of the 28th day, based on the data contained in the medical file and the administrative file.
Over-triage | 28th day
  Over-triage, defined by the management of severely traumatized patients in the trauma centre and whose ISS is less than or equal to 15 and who do not present any of the following criteria :
  * the need for transfusion of more than 4 red blood cell concentrates during the first 6 hours of management;
  * the presence of severe head trauma with CT scan lesions;
  * the presence of a spinal cord injury;
  * the need for specialized emergency surgery (laparotomy or hemostasis thoracotomy, embolization, craniectomy, intracranial pressure measurement, chest drainage) within the first 24 hours;
  * the need for transfer to a trauma center. This variable will be evaluated at the end of the 28th day, based on the data contained in the medical file and in the administrative file
Transfer to a trauma centre | 1 day
  Tranfer to a trauma centre at the end of the pre-hospital phase. This criterion will be evaluated at the time of admission of the patient out of the SMUR ambulance. Trauma centres are considered to be hospitals with a unit dedicated to the care of these patients, identified as such by the territorially competent regional health agency;
Secondary inter-hospital transfer | 28th day
  The need for secondary inter-hospital transfer to a specialized trauma centre or a higher-level trauma centre. This variable is defined as the transfer of the patient, during the study period, from a hospital that does not have a trauma centre to the trauma centre of a hospital that does, or the transfer of the patient from a hospital trauma centre to a higher level trauma centre (III to II, II to I, III to I). This variable will be evaluated at the end of day 28, based on the data contained in the medical file and the administrative file. Transfers for specialized but non-urgent care (e.g. hand microsurgery that can be carried out beyond the first 24 hours) will not be counted as secondary inter-hospital transfers;
Days living without mechanical ventilation | 28th day
  The number of days living without mechanical ventilation during the first 28 days. This criterion will be assessed at the end of the 28th day, by subtracting from 28 the number of days the patient received ventilatory support by mechanical ventilation. The change of day is made at midnight. By definition, deceased patients are assigned 0 days without mechanical ventilation;
Days living without resuscitation | 28th day
  The number of days living without resuscitation during the first 28 days. This criterion will be assessed at the end of the 28th day, by subtracting from 28 the number of days the patient will have been in resuscitation. The change of day is made at midnight. By definition, deceased patients are assigned 0 days out of resuscitation;
Length of stay in resuscitation | 28th day
  This variable will be evaluated at the end of the 28th day, based on the data contained in the medical record and in the administrative file;
Modalities of the post-traumatic injury assessment by chest X-ray | first 24 hours of hospitalization
  This criterion will be assessed at the end of the first 24 hours of hospitalization. It will be assessed by first performing a chest X-ray
Modalities of the post-traumatic injury assessment by pelvis X-ray | first 24 hours of hospitalization
  This criterion will be assessed at the end of the first 24 hours of hospitalization. It will be assessed by first performing a pelvis X-ray
Modalities of the post-traumatic injury assessment by abdominal ultrasound | first 24 hours of hospitalization
  This criterion will be assessed at the end of the first 24 hours of hospitalization. It will be assessed by first performing an abdominal ultrasound
Modalities of the post-traumatic injury assessment by transcranial Doppler scan | first 24 hours of hospitalization
  This criterion will be assessed at the end of the first 24 hours of hospitalization. It will be assessed by first performing a transcranial Doppler scan
Modalities of the post-traumatic injury assessment by CT scan | first 24 hours of hospitalization
  This criterion will be assessed at the end of the first 24 hours of hospitalization. This evaluation will include a whole body CT scan with contrast media injection
Modalities of the post-traumatic injury assessment by bone radiographs | first 24 hours of hospitalization
  This criterion will be assessed at the end of the first 24 hours of hospitalization. This evaluation will include guided bone radiographs;
Need for and timing of laparotomy | 28th day
  The need for and timing of laparotomy within the first 24 hours. This variable will be evaluated at the end of the 28th day, based on the data contained in the medical file and in the administrative file;
Need for and timing of hemostasis thoracotomy | 28th day
  The need for and timing of hemostasis thoracotomy within the first 24 hours. This variable will be evaluated at the end of the 28th day, based on the data contained in the medical file and in the administrative file;
Need for and timing of embolization | 28th day
  The need for and timing of embolization within the first 24 hours. This variable will be evaluated at the end of the 28th day, based on the data contained in the medical file and in the administrative file;
Need for and timing of craniectomy | 28th day
  The need for and timing of craniectomy within the first 24 hours. This variable will be evaluated at the end of the 28th day, based on the data contained in the medical file and in the administrative file;
Need for and timing of intracranial pressure measurement | 28th day
  The need for and timing of intracranial pressure measurement within the first 24 hours. This variable will be evaluated at the end of the 28th day, based on the data contained in the medical file and in the administrative file;
Need for and timing of chest drainage | 28th day
  The need for and timing of chest drainage within the first 24 hours. This variable will be evaluated at the end of the 28th day, based on the data contained in the medical file and in the administrative file;
Distance to the nearest available pre-hospital medical facility | 1 day
  The distance to the nearest available pre-hospital medical facility. This variable is defined as the distance between the accident and the nearest available pre-hospital medical facility (light vehicles, mobile hospital units, helicopters) available at the time of the alert in the department concerned.
Length of mechanical ventilation | 28th day
  This variable will be evaluated at the end of the 28th day, based on the data contained in the medical record and in the administrative file;
Length of hospital stay | 28th day
  This variable will be evaluated at the end of the 28th day, based on the data contained in the medical record and in the administrative file;

CONTACTS AND LOCATIONS:
Overall Officials: RAUX Mathieu, MD PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Pitié-Salpetrière, Paris, France

IPD SHARING:
Plan to Share IPD: No